CLINICAL TRIAL: NCT02429063
Title: Light Therapy to Increase Energy in Adolescents and Young Adults Newly Diagnosed With Solid Tumors: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of California, San Diego (Other); University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LITE; NCI-2015-00679 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Neoplasms; Fatigue
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright White Light (Experimental): Participants use the bright white light intervention for 30 minutes upon waking each morning for 60 days.
  Interventions: Other: Bright White Light
- Dim Red Light (Experimental): Participants use the dim red light intervention for 30 minutes upon waking each morning for 60 days.
  Interventions: Other: Dim Red Light

INTERVENTIONS:
Other: Bright White Light — The light will be administered via a Litebook Elite or Litebook Advantage (Litebook®, Ltd., Medicine Hat, Canada). The Litebook® is a small (6×5×1 in.) and lightweight (8 oz.) box and will be fitted with adherence monitors to record at what time and for what duration the light box is turned on. The Litebook® is designed to be placed on a table approximately 18 inches from the participant's head and within 45° of the midline of the visual field. The BWL Litebook® looks identical to the DRL and utilizes 24 white light-emitting diode (LED) lights and does not emit ultraviolet light.
  Other Names: Litebook®; BWL
  Arms: Bright White Light
Other: Dim Red Light — The light will be administered via a Litebook Elite or Litebook Advantage (Litebook®, Ltd., Medicine Hat, Canada). The Litebook® is a small (6×5×1 in.) and lightweight (8 oz.) box and will be fitted with adherence monitors to record at what time and for what duration the light box is turned on. The Litebook® is designed to be placed on a table approximately 18 inches from the participant's head and within 45° of the midline of the visual field. The DRL Litebook looks identical to the BWL box and contains red lights rather than white LED lights.
  Other Names: Litebook®; DRL
  Arms: Dim Red Light

SUMMARY:
Fatigue is one of the most consistent and distressing symptoms reported by pediatric oncology patients. The investigators' work has demonstrated that in the period from diagnosis through the initial 8 weeks of treatment, adolescents and young adults with solid tumors experience substantial fatigue that is not related to sleep disruption. Fatigue can contribute to many adverse outcomes including poor treatment adherence, reduced social activities, depressive symptoms, behavior problems, and poorer quality of life. Unfortunately, no definitive intervention to reduce fatigue has been developed for pediatric oncology patients. Investigators propose a study to estimate the feasibility and acceptability of bright light therapy as an intervention to decrease fatigue in adolescents and young adults who are newly diagnosed and receiving treatment for solid tumors, including lymphoma.

DETAILED DESCRIPTION:
This feasibility and acceptability study will assess the rate of consent to, adherence to, and side effects from a therapy study in a randomized trial comparing bright white light (BWL) to dim red light (DRL). Four questionnaires will be distributed to patients and/or their parents, depending upon the questionnaire, to study the fatigue, quality of life, mood symptoms, and side effects of the BWL/DRL intervention in adolescents and young adults being treated for solid tumors, including lymphoma.

PRIMARY OBJECTIVES:

* To estimate the feasibility and acceptability of a BWL intervention compared to a DRL standard comparison group in adolescent/young adult solid tumor and lymphoma patients.

SECONDARY OBJECTIVE:

* To estimate the effect size of this intervention on measures of fatigue in order to design a larger clinical trial of efficacy of a randomized control trial of BWL versus DRL intervention for fatigue in pediatric oncology patients.

OTHER PRESPECIFIED OBJECTIVES:

* Estimate the effect of participant location (inpatient, hospital-based housing, or home) on adherence.
* Estimate rates of depressive symptoms.
* Describe quality of life.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 12 years or older
* Has initiated treatment as part of an active St. Jude Children's Research Hospital (SJCRH) treatment plan
* ≤ 30 days post diagnosis of a solid tumor or lymphoma
* Patient speaks, reads and writes in English or Spanish
* Potential participant/guardian is willing to sign informed consent

EXCLUSION CRITERIA:

* Blind or having a history of eye disease including, but not limited to, macular degeneration, or other diagnosed retinal problems
* Undergone laser corrective eye surgery in the past 30 days
* Significant physiological or psychological impairment that interferes with participation (e.g., migraines, bipolar disorder, psychosis, seasonal affective disorder)
* Recently started on anti-depressant medications (past one month for those on Selective Serotonin Reuptake Inhibitors [SSRI] and past two months for those started on Monoamine Oxidase Inhibitors [MAOI])

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Rate of consent | Day 0
  Estimate the rates of consent to a BWL intervention, compared to DRL in adolescent/young adult solid tumor and lymphoma patients.
Rate of adherence | At the end of therapy (Day 60)
  Estimate the rates of adherence to the intervention in adolescent/young adult solid tumor or lymphoma patients for each group.
Rate of side effects | At the end of therapy (Day 60)
  Estimate rates of side effects in a light therapy intervention trial.

SECONDARY OUTCOMES:
Rate of fatigue | At the end of therapy (Day 60)
  Estimate the rates of fatigue between the intervention and comparison groups. Fatigue will be measured by self- and parent-report with the 18-item PedsQL™ Multidimensional Fatigue Scale (MFS) that includes three subscales: (1) general fatigue (six items), (2) sleep/rest fatigue (six items), and (3) cognitive fatigue (six items).

OTHER OUTCOMES:
Rate of adherence by participant location | At the end of therapy (Day 60)
  Estimate the effect of participant location (inpatient, hospital-based housing, or home) on adherence.
Rate of depressive symptoms | Baseline (Day 0), and approximately Day 14, Day 28 Day 42, and Day 60
  Mood symptoms will be assessed with the Children's Depression Inventory, 2nd Edition (CDI 2) in participants 8-17 years old and by the BDI-II in participants 18 years of age and older. The CDI 2 is a 27-item self-report measure of depressive symptoms in children ages 7-17.
Metrics of quality of life and well-being | Baseline (Day 0), and approximately Day 14, Day 28, Day 42, and Day 60
  Quality of life will be assessed by self- and parent-report with the PedsQL™ Acute Version [34] that includes 4 subscales: (1) physical functioning (eight items), (2) emotional functioning (five items), (3) social functioning (five items), and (4) school functioning (five items) as well as a total score. The Likert scale and scoring method are identical to the MFS, with higher scores indicating better health-related quality of life. The PedsQL™ will be completed prior to initiation of the intervention, at three time points during the intervention period (14 +/- 3, 28 +/- 3 days, and 42 +/- 3 days) , and at the end of the 60 day intervention/period (days 61-68).

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Crabtree, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Crabtree VM, LaRosa KN, MacArthur E, Russell K, Wang F, Zhang H, Pan H, Brigden J, Schwartz LE, Wilson M, Pappo A. Feasibility and Acceptability of Light Therapy to Reduce Fatigue in Adolescents and Young Adults Receiving Cancer-Directed Therapy. Behav Sleep Med. 2021 Jul-Aug;19(4):492-504. doi: 10.1080/15402002.2020.1797744. Epub 2020 Aug 4. PMID 32746639
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols